CLINICAL TRIAL: NCT00561366
Title: A Multicenter, Double-Blind, Placebo-Controlled, Phase 2b Study to Investigate the Safety and Efficacy of Arimoclomol in Volunteers With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: A Multicenter, Double-Blind Study to Investigate the Safety and Efficacy of Arimoclomol in Volunteers With ALS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Not moving forward with program.
Sponsor: CytRx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AALS-003
Record Dates: First submitted 2007-11-16; First posted 2007-11-20 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Lou Gehrig's disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — arimoclomol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Experimental)
  Interventions: Drug: Arimoclomol

INTERVENTIONS:
Drug: Placebo — Placebo t.i.d.
  Arms: 1
Drug: Arimoclomol — capsule, 400 mg t.i.d.
  Arms: 2

SUMMARY:
Arimoclomol is a small molecule that upregulates "molecular chaperones" in cells under stress. Arimoclomol extends survival by five weeks when given both pre-symptomatically and at disease onset in a mutant superoxide dismutase (SOD1) transgenic mouse model of ALS. Furthermore, it has been demonstrated to have neuroprotective and neuroregenerative effects in other rat models of nerve damage. Molecular chaperone proteins are critical in the cellular response to stress and protein misfolding. Recent data suggest that the SOD1 mutation responsible for ALS in some patients with familial disease reduces the availability of a variety of molecular chaperones, and thus weakens their ability to respond to cellular stress. Protein misfolding and consequent aggregation may play a role in the pathogenesis of both the familial and sporadic forms of ALS. Therapeutic agents such as arimoclomol that improve cellular chaperone response to protein misfolding may be helpful in ALS.

DETAILED DESCRIPTION:
This is a Phase 2b double-blind, randomized, placebo-controlled parallel-group study evaluating the safety and efficacy of arimoclomol (400 mg t.i.d.) compared to placebo. A safety lead-in phase will be employed to ensure the safety of all study volunteers.

Tier I (Safety Lead-in): During the enrollment period for the safety lead-in phase, 24 volunteers meeting inclusion/exclusion criteria will be randomized at 4 investigative sites. These volunteers will have weekly visits during the first 4 weeks after starting treatment. Pharmacokinetics (PK) will be performed at various timepoints throughout these 4 weeks. After the initial 4 weeks of treatment, visits will continue at 4-week intervals up to Week 36, subsequently visits will occur every 8 weeks up to Week 68. A final visit will occur at Week 72. There will be a 28-day post study medication Follow-Up Telephone Call to assess medical status and adverse events.

Tier II: After the Tier I volunteers finish 4 weeks of treatment, their data will be reviewed by the IDMC and, if no serious safety issues are identified, the recommendation will be made to start the second enrollment period (Tier II). During Tier II enrollment, volunteers recruited from approximately 30 to 40 centers in the US and Canada will be randomized. After screening and randomization, volunteers will be followed every 4 weeks for 9 months. Subsequently visits will occur every 8 weeks up to Week 68, with interim Follow-Up Telephone Calls at Weeks 16, 24, and 32 and a final visit at Week 72. A Week 76 Follow-Up Telephone Call to assess medical status and adverse events will occur at 28 days post last dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

* Familial or sporadic ALS.
* Diagnosed with laboratory-supported probable, probable or definite ALS according to the World Federation of Neurology El Escorial criteria for less than or equal to 36 months' duration prior to the Screening Visit.
* Vital capacity (VC) equal to or greater than 70% predicted value for gender, height and age at the Screening Visit.
* Geographic accessibility to the study site.
* Ability to take oral medication at the Screening Visit, based on verbal report.
* Fluency in English, Spanish or Canadian French.

Exclusion Criteria:

* History of known sensitivity or intolerability to arimoclomol or to any other related compound.
* Prior exposure to arimoclomol through a clinical trial or physician-sponsored IND.
* Exposure to any investigational agent within 30 days of the Screening Visit.
* Presence of any of the following clinical conditions:

  1. Substance abuse within the past year
  2. Unstable cardiac, pulmonary, renal, hepatic, endocrine, hematologic, or active malignancy or infectious disease
  3. AIDS or AIDS-related complex
  4. Unstable psychiatric illness defined as psychosis (hallucinations or delusions), untreated major depression within 90 days of the Screening Visit.
* Laboratory values: Screening serum creatinine greater than or equal to 1.5 mg/dL, creatinine clearance less than 70 cc/min, alanine aminotransferase (ALT) greater than 3.0 times the upper limit of normal, total bilirubin greater than 1.5 times the upper limit of normal, white blood cell (WBC) count less than 3,500/mm3, platelet concentration of <100,000/ul, hematocrit level of less than 33 % for female or less than 35 % for male, or coagulation tests (PT, PTT) greater than or equal to 1.5 times upper limit of normal.
* Female volunteers who are breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
ALSFRS-R | 9 months

SECONDARY OUTCOMES:
ALSFRS-R | 18 months
Survival | 18 months
Muscle strength | 9 and 18 months
Pulmonary function | 9 and 18 months
MUNE | 9 and 18 months
Quality of Life | 9 and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Merit Cudkowicz, MD, MSc, Principal Investigator — Massachusetts General Hospital; Jeremy Shefner, MD, PhD, Principal Investigator — State University of New York - Upstate Medical University
Locations (35):
- United States (31):
  - University of California Los Angeles - Tier 2 Site, Pacific Palisades, California
  - University of California - San Francisco - Tier 2 Site, San Francisco, California
  - University of Colorado Health Sciences Center - Tier 2 Site, Denver, Colorado
  - University of Miami - Tier 2 Site, Miami, Florida
  - Emory University - Tier 2 site, Atlanta, Georgia
  - Northwestern University, Dept. of Neurology - Tier 2 Site, Chicago, Illinois
  - University of Kansas Medical Center - Tier 2 site, Kansas City, Kansas
  - John Hopkins University - Tier 2 Site, Baltimore, Maryland
  - Massachusetts General Hospital - Tier 1 Site, Boston, Massachusetts
  - Baystate Medical Center - Tier 2 Site, Springfield, Massachusetts
  - Saint Louis University, Neuromuscular Div. - Tier 2 Site, St Louis, Missouri
  - Washington University - Tier 2 Site, St Louis, Missouri
  - BryanLGH Medical Center - Tier 2 Site, Lincoln, Nebraska
  - Upstate Clinical Research, LLC - Tier 2 Site, Albany, New York
  - Mount Sinai School of Medicine - Tier 2 Site, New York, New York
  - Columbia University Medical Center - Tier 2 site, New York, New York
  - SUNY Downstate Medical Center - Tier 1 Site, Syracuse, New York
  - Duke University Medical Center - Tier 1 Site, Durham, North Carolina
  - Wake Forest University School of Medicine -Tier 2 Site, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation -Tier 2 site, Cleveland, Ohio
  - Providence ALS Center - Tier 2 Site, Portland, Oregon
  - Pennsylvania State University School of Medicine - Tier 2 Site, Hershey, Pennsylvania
  - Drexel University College of Medicine - Tier 1 Site, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center - Tier 2 Site, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center - Tier 2, Nashville, Tennessee
  - Texas Neurology, PA - Tier 2 Site, Dallas, Texas
  - University of Texas Health Science Center - Tier 2 Site, San Antonio, Texas
  - University of Vermont, College of Medicine - Tier 2, Burlington, Vermont
  - University of Virginia - Tier 2 Sites, Charlottesville, Virginia
  - Virginia Mason Clinic - Tier 2 Site, Seattle, Washington
  - Medical College of Wisconsin - Tier 2 Site, Milwaukee, Wisconsin
- Canada (4):
  - University of British Columbia, Gordon and Leslie Diamond Health Care Centre - Tier 2 Site, Vancouver, British Columbia
  - London Health Science Center - Tier 2 Site, London, Ontario
  - University of Toronto, Sunnybrook Health Sciences Centre - Tier 2 Site, Toronto, Ontario
  - Montreal Neurological Institute - Tier 2, Montreal, Quebec